CLINICAL TRIAL: NCT04344197
Title: Surgery During Covid-19: The Role of Asymptomatic Patients, a Survey
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Associate Professor, Head of Department, University of Rome Tor Vergata
Other Study IDs: s-covid survey
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Surgery; COVID; Asymptomatic Patient; Covid-19; Preventive Measures
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: global survey — surgery questionnaire

SUMMARY:
a brief questionnaire to get a clearer picture of the situation regarding surgical patients with special emphasis on asymptomatic Covid-19 patients.

DETAILED DESCRIPTION:
With new evidence on the role of asymptomatic patients in spreading the disease during the Covid-19 pandemic, symptom driven guidelines for testing, hospital allocation and personal protective equipment (PPE) use do not seem appropriate to limit in-hospital transmission. At time when lockdowns are in place in most countries, hospitals can become the new source of infection.

Guidelines are very variable depending on local policies and availability of medical supplies, resulting in most hospitals taking different preventive measures.

ELIGIBILITY:
Inclusion Criteria:

general surgeon

Exclusion Criteria:

other speciality

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: surgeon
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
overview of surgical management on preventive measures of hospital infection spread during covid 19 | 2/04/2020 to 15/04/2020

SECONDARY OUTCOMES:
testing policies and preventive measures for Covid-19, and their association with asymptomatic cases. | 02/04/2020 to 15/04/2020

CONTACTS AND LOCATIONS:
Locations (1):
- Tor Vergata Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bellato V, Konishi T, Pellino G, An Y, Piciocchi A, Sensi B, Siragusa L, Khanna K, Pirozzi BM, Franceschilli M, Campanelli M, Efetov S, Sica GS; S-COVID Collaborative Group. Screening policies, preventive measures and in-hospital infection of COVID-19 in global surgical practices. J Glob Health. 2020 Dec;10(2):020507. doi: 10.7189/jogh.10.020507. PMID 33110590